CLINICAL TRIAL: NCT02699528
Title: Does Methylphenidate, Prescribed for Attention Deficit Disorder, Influence Primary Enuresis in These Children?
Brief Title: The Effect of Methylphenidate on Primary Enuresis in Children With Attention Deficit Hyperactivity Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Natan Watemberg, MD, Meir Medical Center
Other Study IDs: MMC-15-0329
Record Dates: First submitted 2016-02-02; First posted 2016-03-04 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Attention Deficit Hyperactivity Disorder; Enuresis
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Enuresis | interventions — Methylphenidate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: methylphenidate — The drug will be prescribed as indicated for attention deficit disorder
  Other Names: Ritalin, Concerta

SUMMARY:
To assess wether methylphenidate reduces the prevalence of primary nocturnal enuresis in children with attention deficit disorder

DETAILED DESCRIPTION:
Children aged 5 - 10 years newly diagnosed with attention deficit hyperactivity disorder who report primary nocturnal enuresis, Investigators will obtain baseline data (from parents/caregivers) on their sleep habits and enuresis characteristics by questionnaire. After 6 weeks of methylphenidate therapy, prescribed for the attention deficit, a new questionnaire will be filled.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of attention deficit hyperactivity disorder
* History of primary nocturnal enuresis
* Normal neurological examination

Exclusion Criteria:

* Anatomical abnormality of the genitourinary system
* Concommitant treatment, pharmacological/behavioral for enuresis
* Concommitant diurnal enuresis

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 5 - 10 years receiving a new diagnosis of attention deficit hyperactivity disorder
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
A reduction in nocturnal enuresis frequency | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Watemberg, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No